CLINICAL TRIAL: NCT05692076
Title: The Role of High Velocity Nasal Insufflation in Prevention of Respiratory Complications in Severe Chest Trauma
Brief Title: Role of HVNI in Severe Chest Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Yasser Abdelgaber, Mohamed yasser, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVNI in severe chest trauma
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Chest Trauma
Keywords: High velocity nasal insufflation
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Intervention Model Description: • we sought statistical advice regarding the sample size needed for the study
  sample size was calculated using G power program to detect significant difference.
  * To detect the incidence of atelectasis in these patients we performed a pilot study included 15 patients using simple mask as oxygen therapy, the results showed an incidence of 50% rate of atelectasis according to the inclusion and exclusion criteria
  * To be able to detect 30% reduction in the incidence of atelectasis we need to include 43 patients in each group
  * Alpha error=.05, 80 % power of the study with equal group assignment
  Group (A) :43 patients (control group):
  • Patient will receive conventional oxygen therapy via nasal prongs , normal oxygen mask or venturi mask
  Group (B) 43 patients ( HVNI group):
  • Patient will receive HVNI therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVNI group (Experimental): Patients will receive high velocity nasal insufflation therapy
  Interventions: Device: High Velocity Nasal Insufflation
- Control group (Other): Patient will receive conventional oxygen therapy via nasal prongs , normal oxygen mask or venturi mask
  Interventions: Device: High Velocity Nasal Insufflation

INTERVENTIONS:
Device: High Velocity Nasal Insufflation — High-flow humidified oxygen with flow rates from 30 to100 L/min with high fraction of inspired oxygen( FiO2) is able to be delivered.

SUMMARY:
to compare the respiratory complications in patient managed with high velocity nasal insufflation versus patients managed with conventional low flow oxygen in patients with severe chest trauma

DETAILED DESCRIPTION:
* Chest trauma are associated with significant morbidity and mortality due to respiratory failure and pneumonia.
* The two main goals of therapy are pain management and pulmonary care and support. There is strong evidence for providing good analgesia to facilitate volume expansion treatment and chest physiotherapy, aiming for deep breathing and effective cough to reduce secretions and prevent the atelectasis.
* Oxygen supplementation is often included as supportive therapy added to bundles of care for patients of chest trauma with rib fractures.

High -velocity nasal insufflation (HVNI ) was first developed for neonates and has gained increasing use in adult patients for prevention and treatment of respiratory failure. High-flow humidified oxygen with flow rates from 30 to100 L/min with high fraction of inspired oxygen( FiO2) is able to be delivered. Positive end-expiratory pressure can be generated, preventing alveoli collapse. The washout of carbon dioxide (CO2)and replacement with enriched O2 purportedly decreases work of breathing and increases breathing effectiveness.

* Routine tests for chest injuries include chest X-rays and computed tomography (CT) scans. Ultrasound has the advantages of being inexpensive, readily available and being free of ionizing radiation .
* In thoracic trauma cases, ultrasonography of the lungs is valuable for evaluating various chest diseases, including chest wall haematoma and fractures, pleural cavity involvement with pleural effusion, haemothorax, and pneumothorax. The ultrasound can also assess the reduce in lung aeration by changing the lung surface and generating distinct patterns as in pulmonary contusions and compression atelectasis.

ELIGIBILITY:
Inclusion Criteria:

* Chest trauma patients with lung injury confirmed by ct imaging

  * the age from 15-55 years old
  * No indication of mechanical ventilation at the time of admission to the intensive care unit

Exclusion Criteria:

* • Patients < 15years old

  * requiring endotracheal intubation and mechanical ventilation immediately on admission for any cause
  * facial fractures or base of skull fractures
  * Who did not receive a chest computed tomography (CT) scan
  * Glasgow Coma Scale <10
  * Massive surgical emphysema
  * COPD Patients ( chronic obstructive pulmonary disease )

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of atelectasis in chest trauma patients | 3 years
  Incidence of atelectasis in chest trauma patients using the chest ultrasound measured by lung consolidation score.

SECONDARY OUTCOMES:
respiratory complications,hospital stay and Comfort levels | 3 years
  Other respiratory complications as hypoxemia and pneumonia.
  * Need for intubation and mechanical ventilation
  * Length of ICU and hospital stay.
  * Comfort levels with different levels of oxygen delivery measured by Likert scale.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karim A, Arora VK. Applications of ultrasonography in respiratory intensive care. Indian J Chest Dis Allied Sci. 2014 Jan-Mar;56(1):27-31. PMID 24930204
- [Background] Easter A. Management of patients with multiple rib fractures. Am J Crit Care. 2001 Sep;10(5):320-7; quiz 328-9. PMID 11548565
- [Background] McGillicuddy D, Rosen P. Diagnostic dilemmas and current controversies in blunt chest trauma. Emerg Med Clin North Am. 2007 Aug;25(3):695-711, viii-ix. doi: 10.1016/j.emc.2007.06.004. PMID 17826213
- [Background] Papazian L, Corley A, Hess D, Fraser JF, Frat JP, Guitton C, Jaber S, Maggiore SM, Nava S, Rello J, Ricard JD, Stephan F, Trisolini R, Azoulay E. Use of high-flow nasal cannula oxygenation in ICU adults: a narrative review. Intensive Care Med. 2016 Sep;42(9):1336-49. doi: 10.1007/s00134-016-4277-8. Epub 2016 Mar 11. PMID 26969671
- [Background] Helviz Y, Einav S. A Systematic Review of the High-flow Nasal Cannula for Adult Patients. Crit Care. 2018 Mar 20;22(1):71. doi: 10.1186/s13054-018-1990-4. PMID 29558988
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Abdalla W, Elgendy M, Abdelaziz AA, Ammar MA. Lung ultrasound versus chest radiography for the diagnosis of pneumothorax in critically ill patients: A prospective, single-blind study. Saudi J Anaesth. 2016 Jul-Sep;10(3):265-9. doi: 10.4103/1658-354X.174906. PMID 27375379
- [Background] Wongwaisayawan S, Suwannanon R, Sawatmongkorngul S, Kaewlai R. Emergency Thoracic US: The Essentials. Radiographics. 2016 May-Jun;36(3):640-59. doi: 10.1148/rg.2016150064. Epub 2016 Apr 1. PMID 27035835
- See also: Related Info — https://www.intechopen.com/chapters/44472